CLINICAL TRIAL: NCT02706561
Title: Helping Men Adhere to Sexual Rehabilitation Following Prostate Cancer Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Center for Marital and Sexual Health of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-317
Record Dates: First submitted 2016-03-03; First posted 2016-03-11 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer; Erectile Dysfunction
Keywords: 15-317
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction | interventions — Surveys and Questionnaires; Educational Status

ARMS (2):
- Standard care plus the ACT intervention (ACT-ED) (Experimental): SC + ACT-ED-Group A uses Acceptance and Commitment Therapy (ACT). In this group, men focus on: long-term goals of rehabilitation; acceptance of the frustration related to ED; identifying and overcoming barriers; and committing to an erectile rehabilitation program. All participants will be asked to complete a set of questionnaires (baseline). The participants can complete it using your personal computer, one of MSKCC computers, in-person or over the phone. The questionnaires will take about 45-60 minutes to complete. You will also complete the same set of questionnaires at 6, 12, 18, and 24 months following study entry. In both groups, the participant will receive three in-person sessions or phone (30-45 minutes), six brief telephone sessions (5-10 minutes), and six monthly phone calls (5-10 minutes)
  Interventions: Behavioral: questionnaires; Behavioral: three in-person sessions; Behavioral: monthly phone calls; Behavioral: Acceptance and Commitment Therapy for Erectile Dysfunction (ACT-ED)
- SC plus nurse Enhanced Monitoring and Education (EME) (Experimental): SC + EME-Group B uses enhanced monitoring and education. This group focuses on answering questions about the rehabilitation program, manage technical issues related to injections, and the dose titration of injection medication. Participants in this group will also receive education on the side effects and impact of prostate cancer surgery, and strategies for restarting sexual activity. All participants will be asked to complete a set of questionnaires (baseline). You can complete it using your personal computer, one of MSKCC computers, in-person or over the phone. The questionnaires will take about 45-60 minutes to complete. The participant will also complete the same set of questionnaires at 6, 12, 18, and 24 months following study entry. In both groups, the participant will receive three in-person sessions or phone (30-45 minutes), six brief telephone sessions (5-10 minutes), and six monthly phone calls (5-10 minutes).
  Interventions: Behavioral: questionnaires; Behavioral: three in-person sessions; Behavioral: monthly phone calls; Behavioral: Enhanced Monitoring and Education (EME)

INTERVENTIONS:
Behavioral: questionnaires
Behavioral: three in-person sessions
Behavioral: monthly phone calls
Behavioral: Acceptance and Commitment Therapy for Erectile Dysfunction (ACT-ED)
  Arms: Standard care plus the ACT intervention (ACT-ED)
Behavioral: Enhanced Monitoring and Education (EME)
  Arms: SC plus nurse Enhanced Monitoring and Education (EME)

SUMMARY:
The purpose of this study is to test two different ways to help men with sexual rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* As per medical record, early stage prostate cancer (Pathologic Stage 1/2 with Gleason score </=8; or Pathologic Stage 3 with Gleason score =/< 7)
* As per medical record, radical prostatectomy (RP) conducted either at MSKCC or at another institution
* As per medical record, ≤ 9 months post-RP
* As per medical record, moderate erectile functioning pre-surgery (i.e., 15 or greater on the IIEF Erectile Function Domain (EFD) score, or graded their erections as a 1 or 2 on the standard 5 point Urology Erectile Function scale, or have a score of 6 or greater on the 1-10 pre-surgery erectile function scale on the SMRP assessment or have a total score of 15 or greater on items 2-7 on the Prostrate Quality of Life Survey: Sexual Domain)
* As per self report or as per medical record starting penile injections as part of the erectile rehabilitation program at MSKCC
* In the judgment of the consenting professional able to communicate, comprehend, and complete questionnaires in English

Exclusion Criteria:

* Both cavernous nerves fully resected as per surgery report (nerve sparing score of 8 in MSKCC surgeon note), or documented in the progress note that the nerves were fully resected.
* Currently on or has a history of being an Androgen Deprivation Therapy (ADT)
* Has any indication of Prostate-Specific Antigen (PSA)
* As per self report, specific injection phobia
* In the judgment of the consenting professional is unable to provide informed consent and complete study sessions and assessment.
* As per self report or as documented in the medical record, current untreated (e.g. no medication no therapy) major psychiatric disorder (schizophrenia, major depression). Patients diagnosed with a major psychiatric disorder will be reviewed by the study PI to determine eligibility prior to consent.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2015-12-08; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
percentages of patients having an Erectile Function Domain (EFD) total score >= 24 | 1 year
  The EFD score of >= 24 will be used to indicate "good" erectile function. This is both a face valid cut-off, and a cut off that is commonly used in the literature as "good" erectile function following radical prostatectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Nelson, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/